CLINICAL TRIAL: NCT02973607
Title: Effects of a Reduction in Renal Function on Cardiovascular Structure and Function: A 5 Year Study of Kidney Donors.
Brief Title: Effects of a Reduction in Renal Function on Cardiovascular Structure and Function
Acronym: CRIB-DONOR II
Status: Completed | Type: Observational
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Anna Price, Principal Investigator, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: RRK5913
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2018-10

CONDITIONS: Chronic Kidney Disease; Hypertrophy, Left Ventricular; Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertrophy, Left Ventricular; Hypertension | interventions — Nephrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Serum, plasma, acellular urine and DNA (for telomere length).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Donors: Patients who donated a kidney and took part in the original CRIB-DONOR study.
  Interventions: Procedure: Nephrectomy
- Controls: Healthy subjects who took part in the original CRIB-DONOR study.

INTERVENTIONS:
Procedure: Nephrectomy — This is observational in design.
  Groups: Donors

SUMMARY:
Chronic kidney disease (CKD) is present in 1 in 7 of the population and confers a high risk of cardiovascular disease. The pathophysiology of cardiovascular disease in CKD is poorly understood because CKD is always accompanied by confounding factors including the underlying disease process (e.g. diabetes mellitus, systemic vasculitis) and the consequences of CKD including hypertension, anaemia and inflammation.

Nephrectomy in kidney donors causes a 30% reduction in renal function providing an ideal study population to measure prospectively the effects of reduced kidney function on the cardiovascular system.

The CRIB-Donor study (ClinicalTrials.gov Identifier:NCT01028703) demonstrated adverse effects on cardiovascular structure and function at 12 months compared to controls including an increase in left ventricular mass. This proposal will measure the changes in cardiovascular structure and function, cardiovascular age and biochemical changes at 5 years providing information on the long term effects of reduced renal function.

DETAILED DESCRIPTION:
A reduction in renal function at one year in kidney donors is associated with adverse cardiovascular structural and functional changes. Increases in LV mass and perhaps fibrosis along with increased arterial stiffness are associated with adverse changes in prognostic imaging biomarkers and may in the long term contribute to the development of clinical disease such as heart failure and arrhythmia.

It is important to follow this valuable and well characterised cohort of subjects to investigate the further natural history of these cardiovascular effects and determine whether such changes tend to regress, stabilise or worsen over time.

Hypotheses:

The reduction in GFR occurring after surgical uni-nephrectomy in donors is associated with long term adverse cardiac and vascular effects which include:

1. A sustained increased in left ventricular mass, impaired left ventricular systolic and diastolic function and increased left ventricular interstitial fibrosis.
2. Reduced aortic distensibility.
3. Increased systolic but not diastolic blood pressure.
4. Increases in oxidative stress, inflammation and collagen turnover
5. Cardiovascular ageing as evidenced by adverse effects on telomere length and DNA damage.

Study design:

We aim to follow up all 124 patients who originally took part in the CRIB-DONOR study at 5 years and eventually 10 years post nephrectomy.

Statistics and sample size:

Using the effect sizes and variances from our previous work (change in LV mass 7g, SD of change 10g) we calculate that by studying 50 subjects in each group we will have 93% power to detect a difference in LV mass of 7g with an alpha value of 0.05. Due to the nature of a follow up study some drop out can be expected. A minimum of 34 patients is required in each group in order to achieve an 80% power. This effect is clinically important; a fall in LV mass index of one SD has been shown to be associated with a 38% reduction in cardiovascular mortality.

With respect to telomere shortening, assuming mean and SD of base pair length of 5500 and 530 the study will be able to detect a difference of 0.612 SD, i.e. 324 base pairs. A sample size of 50 patients per group would provide a 85% power to detect a difference.

ELIGIBILITY:
Inclusion Criteria:

All patients who took part in the original CRIB-Donor study.

Exclusion Criteria:

Pregnant women

Patients will have previously met nationally set criteria for living donation which excludes those with:

Diabetes mellitus Atrial fibrillation Left ventricular dysfunction (ejection fraction <40% on transthoracic echocardiography) History of cardiovascular or pulmonary disease Evidence of hypertensive end-organ damage.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Living donors and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Left ventricular mass and interstitial fibrosis | 3 years
  Measured by CMR (part 1 of study).

SECONDARY OUTCOMES:
Aortic compliance | 3 years
  Measured by CMR (part 1 of study).
Cardiovascular age | 3 years
  Measured by telomere length and studies of DNA damage (part 1 and 2 of study).
Oxidative stress, inflammation and collagen turnover | 3 years
  Measured by assay and bioassay (part 1 of study).
Blood pressure | 3 years
  Measured by ambulatory blood pressure monitoring (part 1 of study).

CONTACTS AND LOCATIONS:
Overall Officials: Professor John Townend, MbChB, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (1):
- Queen Elizabeth Hospital Birmingham, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No